CLINICAL TRIAL: NCT03131817
Title: Cortical Stimulation to Treat Mood and Behavioral Symptoms in Parkinson's
Brief Title: Cortical Stimulation to Treat Mood and Behavioral Symptoms in Parkinson's Disease Patients
Acronym: PC+S_PFC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Simon J. Little, MBBS, PhD (Other)
Responsible Party: Sponsor-Investigator, Simon J. Little, MBBS, PhD, Assistant Professor, Clinical Neurology, University of California, San Francisco
Organization: University of California, San Francisco (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16-20284
Record Dates: First submitted 2016-09-28; First posted 2017-04-27 (Actual); Results first posted 2025-11-21 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Electric Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Chronic Neural Recording with Prefrontal Cortex ECoG in Parkinson's Disease (Experimental): Participants with Parkinson's disease underwent deep brain stimulation (DBS) lead implantation targeting either the subthalamic nucleus or globus pallidus internus for motor symptom management. A permanent 4-contact subdural electrocorticography (ECoG) strip was also placed over the right prefrontal cortex and connected to a Medtronic Activa PC+S neurostimulator. This setup enabled chronic recording of local field potentials from the prefrontal cortex during daily life and structured experimental tasks.
  Neural and behavioral data were collected through decision-making tasks and longitudinal self-report of mood and symptoms using a tablet-based tool. Clinical DBS and medication adjustments were performed solely as part of standard care and were not influenced by participation in the study.
  Interventions: Device: Medtronic Activa PC+S System with Chronic Neural Recording; Behavioral: Effort-Reward Decision-Making Task; Behavioral: Tablet-Based Mood Tracking (Immediate Mood Scaler)
- Prefrontal Cortex ECoG Stimulation in Parkinson's Disease (Experimental): A subset of participants in the recording cohort also received experimental stimulation through the implanted prefrontal ECoG strip. One participant underwent blinded, block-wise prefrontal cortex stimulation during a behavioral task to assess its causal effects on motivation and decision-making. Additionally, two participants received blinded, chronic prefrontal stimulation at home over a 14-day period, in conjunction with their ongoing subcortical motor DBS. These participants completed daily self-reports of mood and anxiety symptoms during the stimulation period.
  All stimulation protocols were experimental and distinct from routine motor DBS programming. Clinical DBS and medication adjustments were made exclusively as part of routine care and were not affected by the study procedures.
  Interventions: Device: Medtronic Activa PC+S System with Chronic Neural Recording; Behavioral: Effort-Reward Decision-Making Task; Other: Prefrontal Cortex Stimulation; Behavioral: Tablet-Based Mood Tracking (Immediate Mood Scaler)

INTERVENTIONS:
Device: Medtronic Activa PC+S System with Chronic Neural Recording — Participants received a Medtronic Activa PC+S system incorporating standard-of-care DBS leads implanted in the basal ganglia (subthalamic nucleus or globus pallidus internus) for management of Parkinson's disease motor symptoms. Additionally, a permanent 4-contact subdural electrocorticography (ECoG) strip was implanted over the prefrontal cortex (e.g., dorsolateral, orbitofrontal, or frontopolar regions) to enable chronic recording of local field potentials. The system allowed for long-term, wireless neural recordings in naturalistic or task-based conditions.
Behavioral: Effort-Reward Decision-Making Task — Participants performed a structured task involving repeated choices to accept or reject offers requiring different levels of physical effort in exchange for variable rewards. The task was used to assess motivation and effort-based valuation processes.
Other: Prefrontal Cortex Stimulation — In one participant, high-frequency stimulation was delivered to the prefrontal cortex via the ECoG strip during a behavioral paradigm. Stimulation was alternated On and Off in a blinded block-wise fashion during the behavioral task to assess causal effects on motivated behavior. In two patients, orbitofrontal cortex (OFC) stimulation was also assessed chronically at home in a within subject, repeated design.
  Other Names: Electrical Stimulation
  Arms: Prefrontal Cortex ECoG Stimulation in Parkinson's Disease
Behavioral: Tablet-Based Mood Tracking (Immediate Mood Scaler) — Participants used a tablet-based Immediate Mood Scaler (IMS) to self-report symptoms related to depression and anxiety in real-time, naturalistic settings. These repeated, in-the-moment assessments were temporally paired with prefrontal cortical recordings to study physio markers of mood fluctuations over several months. No stimulation was delivered through the prefrontal cortex electrode.

SUMMARY:
This study will investigate cortical stimulation to treat mood and behavioral symptoms in Parkinson's disease patients.

DETAILED DESCRIPTION:
Depression, anxiety and impulse control disorders are among the most prominent neuropsychiatric symptoms in Parkinson's disease (PD) that greatly impact patients' and caregivers' quality of life. However, the neural correlate underlying these symptoms is still largely unknown preventing the development of comprehensive treatment for these symptoms.

The aims of this study are to 1) Determine the neural correlates of non-motor symptoms, 2) Determine how cortical stimulation can reduce these symptoms and normalize the abnormal brain signals, and 3) Teach patients how to voluntarily modulate the abnormal brain signals.

Ten PD patients undergoing deep brain surgery (DBS) implantation and diagnosed with mild to moderate mood disorder and/or impulsive behavior will be enrolled in this study. In addition to the standard therapeutic DBS electrode used to treat motor symptoms, a flexible electrode will be placed over the prefrontal cortex. Both electrodes will be attached to the Medtronic Activa PC+S pulse generator (and Medtronic Summit RC+S pulse generator as replacements), investigational devices that allows therapeutic stimulation and chronic brain recordings. At multiple time points, up to 2 years post-implantation, in our clinic or patient's home, brain signals will be recorded while patients are resting or performing emotion/cognition tasks. Symptoms will be assessed using validated questionnaires and tasks to allow identification of neurophysiological correlates of non-motor symptoms. There is also an optional sleep study included for better understanding of the brain's physiology. The investigators will then investigate the effect of cortical stimulation on both symptoms severity and brain signals that may be related to symptom expression. These signals will then be used to implement closed-loop controlled cortical stimulation and neuro-feedback controlled strategies.

ELIGIBILITY:
Inclusion Criteria:

* Ability to give informed consent for the study
* Age 30-75
* Diagnosis of Parkinson's disease by a movement disorders specialist
* Movement disorder symptoms that are sufficiently severe, in the setting of best medical therapy, to warrant surgical implantation of deep brain stimulators according to standard clinical criteria
* UPDRS-III score off medication between 20 and 80 and an improvement of at least 30% in the baseline UPDRS-III on medication score, compared to the baseline off-medication score.

OR Patients with tremor-dominant PD (a tremor score of at least 2 on a UPDRS-III sub-score for tremor), treatment resistant, with significant functional disability despite maximal medical management OR Patients intolerant to medication causing significant functional disability

* Have one or several mild to moderate mood or impulsive behavior as defined by:

  1. depression (BDI>=13)
  2. anxiety (BAI >=7)
  3. impulsive behavior as indicated by a positive score on the Questionnaire for Impulsive-Compulsive disorders in Parkinson's Disease (QUIP-A) or as determined by clinical interview or informant report
  4. Mood or behavior symptom fluctuations corresponding to minimum 30% improvement in non-motor symptoms when comparing visual analogue scales (VAS) scores in the on versus off medication state
* Stable doses of anti-Parkinsonian medications for at least 30 days prior to their baseline assessment.

Exclusion Criteria:

* Pregnancy or breast feeding
* MRI showing cortical atrophy out of proportion to age
* MRI showing focal brain lesions that could indicate a disorder other than idiopathic PD
* Major comorbidity increasing the risk of surgery (prior stroke, severe hypertension, severe diabetes, or need for chronic anticoagulation other than aspirin)
* Any prior intracranial surgery except DBS surgery
* Significant cognitive impairment (MoCA<20).
* History of seizures
* Immunocompromised
* Has an active infection
* Requires diathermy, electroconvulsive therapy (ECT) or transcranial magnetic stimulation (TMS) to treat a chronic condition
* Inability to comply with study follow-up visits
* Any personality or mood symptoms that study personnel believe will interfere with study requirements.

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2016-12-16 (Actual); Primary Completion 2024-06-18 (Actual); Study Completion 2024-06-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Simon Little, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- UCSF Surgical Movement Disorders Center, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Chronic Neural Recording With Prefrontal Cortex ECoG in Parkinson's Disease: Participants with Parkinson's disease underwent implantation of deep brain stimulation (DBS) leads targeting the basal ganglia (subthalamic nucleus or globus pallidus internus) for motor symptom management, along with a permanent 4-contact subdural electrocorticography (ECoG) strip placed over the right prefrontal cortex. The ECoG strip was connected to a Medtronic Activa PC+S neurostimulator to enable chronic recording of local field potentials from the prefrontal cortex during everyday life and experimental tasks. All participants contributed neural and behavioral data, either during structured decision-making tasks or through longitudinal self-tracking of mood and symptoms using a tablet-based tool. One participant also underwent blinded, block-wise prefrontal cortex stimulation via the ECoG strip during a behavioral task to assess causal effects on motivation and decision-making. Two patients tested at home blinded chronic Prefrontal stimulation over 14 days in addition to their subcortical motor stimulation and provided self report ratings of mood and anxiety. Clinical DBS and medication adjustments were made only as part of routine care and not influenced by study participation.
Period: Overall Study
Arm/Group | Chronic Neural Recording With Prefrontal Cortex ECoG in Parkinson's Disease
Started | 5
Enrollment and Implantation (Five participants with Parkinson's disease who met inclusion criteria (diagnosis of PD, indication for DBS, comorbid mild-to-moderate depression and/or anxiety, and no significant cognitive impairment) were enrolled and underwent surgical implantation of both basal ganglia DBS and a prefrontal cortex ECoG lead.) | 5
Completed (All five implanted participants entered the multi-month chronic recording period pairing ECoG data collection with self-rated mood assessments. One participant developed cognitive decline and was unable to provide regular symptom assessments and was excluded from final analysis.) | 4
Not Completed | 1
Not completed — Participant developed cognitive decline and was unable to provide regular symptom assessments | 1

BASELINE CHARACTERISTICS:
Population: Five participants were enrolled in the study. However, one participant developed cognitive decline during the study and was unable to provide regular symptom assessments, so only four participants were included in the final analysis.
Arm/Group | Chronic Neural Recording With Prefrontal Cortex ECoG in Parkinson's Disease
Number analyzed (Participants) | 4
Age, Categorical [Count of Participants; unit: Participants] — Population: One participant developed cognitive decline and was unable to provide regular symptom assessments and was excluded from final analysis.
  Participants
    <=18 years | 0
    Between 18 and 65 years | 2
    >=65 years | 2
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: One participant developed cognitive decline and was unable to provide regular symptom assessments and was excluded from final analysis.
  years | 61 (7)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: One participant developed cognitive decline and was unable to provide regular symptom assessments and was excluded from final analysis.
  Participants
    Female | 3
    Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: One participant developed cognitive decline and was unable to provide regular symptom assessments and was excluded from final analysis.
  Participants
    Hispanic or Latino | 0
    Not Hispanic or Latino | 4
    Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: One participant developed cognitive decline and was unable to provide regular symptom assessments and was excluded from final analysis.
  Participants
    American Indian or Alaska Native | 0
    Asian | 1
    Native Hawaiian or Other Pacific Islander | 0
    Black or African American | 0
    White | 2
    More than one race | 0
    Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants] — Population: One participant developed cognitive decline and was unable to provide regular symptom assessments and was excluded from final analysis.
  participants
    United States | 4

OUTCOME MEASURES:

1. Primary Outcome: Association Between Basal Ganglia Beta Power and Effort Level (Beta Coefficient)
Description: Mean beta-band (12-20 Hz) oscillatory power in the basal ganglia (BG) during the decision period, analyzed as a function of the current trial effort level during the reward-effort decision-making task.
Time Frame: Single recording session per participant (approximately 90 minutes total; 3 blocks of 25 trials each), with outcome assessed at each trial and data aggregated across all trials for all participants.
Population: as for baseline characteristics
Measure: Number; unit: beta coefficient
Arm/Group | Chronic Neural Recording With Prefrontal Cortex ECoG in Parkinson's Disease
Number analyzed (Participants) | 4
beta coefficient | -0.175
Statistical Analysis 1: Comparison: Chronic Neural Recording With Prefrontal Cortex ECoG in Parkinson's Disease; Test type: Other; p = 0.007, Mixed Models Analysis

2. Primary Outcome: Prefrontal Cortex Theta Power Relative to Previous Trial Reward (Beta Coefficient)
Description: Mean theta-band (4-7 Hz) oscillatory power in the prefrontal cortex (PFC) was assessed during the decision period of each trial. Theta power was modeled as a function of the reward received in the previous trial using linear mixed-effects models. The analysis included trials from structured decision-making task sessions.
Time Frame: as for outcome 1
Population: as for baseline characteristics
Measure: Number; unit: beta coefficient
Arm/Group | Chronic Neural Recording With Prefrontal Cortex ECoG in Parkinson's Disease
Number analyzed (Participants) | 4
beta coefficient | 0.424
Statistical Analysis 1: Comparison: Chronic Neural Recording With Prefrontal Cortex ECoG in Parkinson's Disease; Test type: Other; p = 0.018, Mixed Models Analysis

3. Primary Outcome: Effect of Reward Magnitude and Effort Cost on Offer Acceptance Probability
Description: This outcome measures the effect of reward magnitude and effort cost on the probability of participants accepting offers during a decision-making task. Effects were assessed using generalized linear mixed models (LMMs) to estimate the relationship between reward, effort, and choice behavior.
Time Frame: as for outcome 1
Population: as for baseline characteristics
Measure: Number; unit: beta coefficient
Arm/Group | Chronic Neural Recording With Prefrontal Cortex ECoG in Parkinson's Disease
Number analyzed (Participants) | 4
beta coefficient
  Reward magnitude effect (higher reward, higher acceptance) | 1.05
  Effort cost effect (higher effort, lower acceptance) | -2.37
Statistical Analysis 1: Comparison: Chronic Neural Recording With Prefrontal Cortex ECoG in Parkinson's Disease; This statistical analysis corresponds to the first outcome row, "Reward magnitude effect (higher reward, higher acceptance)." The generalized linear mixed model examined the effect of reward magnitude on the probability of accepting offers; Test type: Other; p < 0.0001, Mixed Models Analysis
Statistical Analysis 2: Comparison: Chronic Neural Recording With Prefrontal Cortex ECoG in Parkinson's Disease; This statistical analysis corresponds to the second outcome row, "Effort cost effect (higher effort, lower acceptance)." The generalized linear mixed model examined the effect of effort cost on the probability of accepting offers; Test type: Other; p < 0.0001, Mixed Models Analysis

4. Primary Outcome: Association Between Prefrontal Cortex Beta Band Spectral Power and Mood Symptoms
Description: This outcome measures the association between prefrontal cortex (PFC) beta band spectral power recorded via chronic subdural ECoG and self-reported symptoms of depression and anxiety assessed using standardized scales. Associations were evaluated using Spearman correlation coefficients calculated for each participant. The Beck Depression Inventory (BDI) ranges from 0 to 63, with higher scores indicating more severe depressive symptoms. The Beck Anxiety Inventory (BAI) ranges from 0 to 63, with higher scores indicating more severe anxiety symptoms.
Time Frame: Daily paired assessments of neural recordings and IMS scores over 3-5 months for each participant.
Population: as for baseline characteristics
Measure: Median (Full Range); unit: Spearman correlation coefficient (r)
Arm/Group | Chronic Neural Recording With Prefrontal Cortex ECoG in Parkinson's Disease
Number analyzed (Participants) | 4
Spearman correlation coefficient (r) | 0.415 [0.31 to 0.48]

5. Primary Outcome: Effect of Chronic Orbitofrontal Cortex (OFC) Stimulation on Depression, Anxiety, and Energy Ratings
Description: This outcome measures self-reported symptoms of depression, anxiety, and energy levels in participants undergoing chronic orbitofrontal cortex (OFC) stimulation at home. Participants received blinded OFC stimulation for 14 days, with alternating sham and active stimulation days. Symptoms were assessed daily using visual analogue scales (VAS) for depression, anxiety, and energy, as well as the Hamilton Depression Rating Scale (HAM-D). The VAS ranges from 0 to 100. For the depression and anxiety VAS, higher scores indicate worse symptoms, whereas for the energy VAS, higher scores indicate greater energy. The HAM-D ranges from 0 to 52, with higher scores indicating more severe depressive symptoms.
Time Frame: Daily paired assessments of neural recordings and IMS scores over 14 days for each participant.
Population: Five participants were enrolled in the study. 2 participants completed this (1 participant dropped out of research activities, 1 declined and 1 moved away from the study centre and so couldn't be followed).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Chronic Neural Recording With Prefrontal Cortex ECoG in Parkinson's Disease
Number analyzed (Participants) | 2
score on a scale
  VAS Anxiety Score (Sham Condition) | 23.23 (23.71)
  VAS Energy Score (Sham Condition) | 67.62 (23.59)
  VAS Depression Score (Sham Condition) | 19.15 (22.71)
  VAS Anxiety Score (Active Condition) | 33.00 (30.35)
  VAS Energy Score (Active Condition) | 71.06 (20.24)
  VAS Depression Score (Active Condition) | 28.63 (28.45)
  HAM-D Score (Sham Condition) | 2.31 (2.72)
  HAM-D Score (Active Condition) | 2.25 (2.96)

6. Secondary Outcome: Effect of Prefrontal Cortex Stimulation on Acceptance Rate of Work Offers During Effort-Based Decision-Making Task
Description: Measured the effect of high-frequency prefrontal cortex (PFC) stimulation on the acceptance rate of work offers during an effort-based decision-making task in one participant (PD5). Stimulation was delivered in a single-blinded, randomized, counterbalanced block-wise design at an amplitude below detectability threshold and without motor effects. Acceptance rate was modeled using a linear mixed model with stimulation condition (On vs Off) as a fixed effect.
Time Frame: Six recording blocks (three with stimulation On and three with stimulation Off), each approximately 15 minutes in duration (total ~90 minutes), with outcome assessed on each trial and data aggregated across both conditions for the participant.
Population: One participant performed the decision-making task with PFC stimulation alternated On and Off between blocks.
Measure: Number; unit: beta coefficient
Arm/Group | Chronic Neural Recording With Prefrontal Cortex ECoG in Parkinson's Disease
Number analyzed (Participants) | 1
beta coefficient | 9.646

ADVERSE EVENTS:
Time Frame: From enrollment until study exit (defined as device explantation or study withdrawal), up to 7 years.
Arm/Group | Chronic Neural Recording With Prefrontal Cortex ECoG in Parkinson's Disease
All-Cause Mortality (participants affected / at risk) | 0/5
Serious Adverse Events (participants affected / at risk) | 2/5
Other Adverse Events (participants affected / at risk) | 1/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Chronic Neural Recording With Prefrontal Cortex ECoG in Parkinson's Disease (N=5)
DBS lead migration requiring repositioning surgery (Injury, poisoning and procedural complications) | 1 (1) — Lead migrated 16mm; patient returned to OR on post-op day 3 for 40-minute repositioning surgery
Prolonged hospitalization with cognitive and executive dysfunction (General disorders) | 1 (3) — Hospitalization prolonged by 6 days post-surgery due to lethargy and confusion; patient later experienced cognitive decline and executive dysfunction possibly related to initial event, managed with medication changes.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Chronic Neural Recording With Prefrontal Cortex ECoG in Parkinson's Disease (N=5)
Cortical lead migration detected post-surgery (Injury, poisoning and procedural complications) | 1 (1) — X-ray 2 months post-surgery showed lead migration; subsequent imaging confirmed no further movement through Oct 2017

LIMITATIONS AND CAVEATS:
The study was limited by a small sample size (n=5) and the absence of a control group. PFC stimulation was tested in only one (in laboratory testing) or two (at-home testing) participants per paradigm due to participant preference and availability. Stimulation was restricted to the right PFC, and recordings were localized to specific basal ganglia and PFC regions. Larger, controlled studies with more diverse samples are needed to address these limitations.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-08-20): https://cdn.clinicaltrials.gov/large-docs/17/NCT03131817/Prot_SAP_000.pdf